CLINICAL TRIAL: NCT01892514
Title: Combined Treatment of Early and Advanced Osteonecrosis of the Femoral Head With Core Decompression and Grafting With Demineralized Bone Matrix (DBM) or Homologous Lyophilized Bone Chips (LBC) Together With Platelet-rich-fibrin (PRF) and Concentrated Bone Marrow (CBM)
Brief Title: Randomized Clinical Trial for the Treatment of Osteonecrosis of the Femoral Head
Acronym: AVN-13
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVN-13
Record Dates: First submitted 2013-06-25; First posted 2013-07-04 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Osteonecrosis
Keywords: osteonecrosis; bone marrow concentrate; demineralized bone matrix; homologous lyophilized bone chips; autologous platelet rich fibrin; mesenchymal stromal cells
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Demineralized Bone Marrow (DBM) (Experimental): core decompression of necrotic area and graft with a biological product based on Demineralized Bone Matrix (DBM), Platelet-Rich-Fibrin (PRF) and Concentrated Bone Marrow (CBM)
  Interventions: Procedure: core decompression
- Lyophilized Bone Chips (LBC) (Experimental): core decompression of the necrotic area and graft with a biological product based on homologous Lyophilized Bone Chips (LBC), Platelet-Rich Fibrin (PRF) and Concentrated Bone Marrow (CBM)
  Interventions: Procedure: core decompression

INTERVENTIONS:
Procedure: core decompression — core decompression of necrotic area and graft with Platelet-Rich Fibrin (PRF) and Concentrated Bone Marrow (CBM)

SUMMARY:
Femoral head avascular necrosis is a relatively common disease (10,000 - 20,000 yearly new United States of America cases) characterized by ischemic cell necrosis in a hip proximal epiphysis area frequently requiring total Hip Arthroplasty (THA).

Even though THA resolves symptoms and restores good joint function, young patients are prone to major disabilities and require prosthesis revision surgeries.

In this clinical trial a comparison between two groups of patients, treated with the same procedure but with two different regenerative techniques, will be performed:

1. 52 patients with necrosis in an early stage, without deformity of the femoral epiphysis (stage 2A-B-C in Association for Research on Osseous Circulation (ARCO) classification, will undergo wide decompression of the necrotic area and reconstruction with homologous Lyophilized Bone Chips (LBC), growth factors from platelet concentrate Platelet-Rich Fibrin (PRF) and Concentrated Bone Marrow (CBM).
2. 52 patients with necrosis of similar features, without deformity of the femoral epiphysis, will undergo wide decompression of the necrotic area and reconstruction with Demineralized Bone Matrix (DBM), growth factors from Platelet-Rich-Fibrin (PRF) and Concentrated Bone Marrow (CBM).

Patients will be evaluated post-surgery at 6 weeks, 3, 6, 12, and 24 months to assess joint damage evolution by ARCO classification, and hip function by clinical scores (Harris Hip Score (HHS), Western Ontario and McMaster Universities Arthritis Index (WOMAC) Score, and Visual Analogic Scale (VAS)).

DETAILED DESCRIPTION:
Rationale. In vitro study and animal models have shown that Mesenchymal Stromal Cells (MSC) have the capacity to differentiate into osteoblastic lineage and that platelet reach fibrin can represent a clinical source of growth factors, able to accelerate the processes of tissue repair. This study intend to highlight how these factors, associated to two different preparations of bone allograft, may accelerate the formation of new host bone in patients with osteonecrosis of the femoral head that represents a common condition in clinical practice with an high socio-economic impact.

Primary objective of the study is to delay or avoid total hip replacement in patients with early necrosis of the femoral head, using different methods of regenerative medicine.

Secondary end points are described below:

* To assess differences in outcome related to features, etiology and localization of the necrosis of the femoral head and to assess variation in post-operative return to daily activities.
* To characterize the osteogenetic and angiogenic potential of marrow-derived Mesenchymal Stromal Cells (MSC) in patients with avascular necrosis of the femoral head, and to correlate these features with medical history and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with necrosis of the femoral head without fracture of the subchondral bone and without flattening of the head itself (according to ARCO classification 2A, B, C).
* Age between 18 and 60 years.
* Any etiology
* Patients who had undergone a previous orthopaedic treatment for traumatology interventions

Exclusion Criteria:

* Patients under the age of 18 years or more than 60 years.
* Patients not able to provide informed consent to treatment.
* Patients suffering from apparent local infective processes.
* Patients with active neoplastic diseases.
* Patients with necrosis of the femoral head of advanced stages (ARCO 3A, B, C, 4).
* Pregnant patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2013-04 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Reduction of the total necrotic area by Magnetic Resonance Imaging (MRI) | baseline, and 12 months after surgery

SECONDARY OUTCOMES:
Pain reduction by measurement of the Visual Analog Scale (VAS) | baseline, and 6 weeks, 3, 6, 12, 24 months after surgery
Functional status evaluated by Harris Hip Score (HHS) and Western Ontario McMaster Universities Arthritis Index (WOMAC) | baseline, and 6, 12, 24 months after surgery
maintenance of structural integrity of the joint by Radiography (RX) | baseline, and 6 weeks, 3, 6, 12, 24 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dante Dallari, Surgeon, Principal Investigator — Rizzoli Orthopaedic Institute
Locations (3):
- Italy (3):
  - 3rd Orthopaedic and Traumatologic Clinic, prevalently oncologic, Rizzoli Orthopaedic Institute, Bologna
  - S.S.D. Conservative Orthopaedic Surgery and Innovative Techniques, Rizzoli Orthopaedic Institute, Bologna
  - Orthopaedic and Traumatologic Department Policlinico di Modena, Modena

REFERENCES:
- [Background] Dallari D, Fini M, Stagni C, Torricelli P, Nicoli Aldini N, Giavaresi G, Cenni E, Baldini N, Cenacchi A, Bassi A, Giardino R, Fornasari PM, Giunti A. In vivo study on the healing of bone defects treated with bone marrow stromal cells, platelet-rich plasma, and freeze-dried bone allografts, alone and in combination. J Orthop Res. 2006 May;24(5):877-88. doi: 10.1002/jor.20112. PMID 16609976
- [Background] Dallari D, Savarino L, Stagni C, Cenni E, Cenacchi A, Fornasari PM, Albisinni U, Rimondi E, Baldini N, Giunti A. Enhanced tibial osteotomy healing with use of bone grafts supplemented with platelet gel or platelet gel and bone marrow stromal cells. J Bone Joint Surg Am. 2007 Nov;89(11):2413-20. doi: 10.2106/JBJS.F.01026. PMID 17974883